CLINICAL TRIAL: NCT01307254
Title: (BAFLA- Barzilai Fatty Liver and Iron Metabolism Study)
Brief Title: Association Between Non-alcoholic Fatty Liver Disease and Iron Status
Acronym: BAFLA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ornit Cohen (Other)
Collaborators: Prof Doron Zamir (Unknown)
Responsible Party: Sponsor-Investigator, Ornit Cohen, r&d unit, Barzilai Medical Center
Organization: Barzilai Medical Center (Other)
Other Study IDs: BAFLA
Record Dates: First submitted 2011-01-05; First posted 2011-03-02 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: NAFLD - Non Alcoholic Fatty Liver Disease
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non alcoholic fatty liver disease
  Interventions: Procedure: blood analysis
- control
  Interventions: Procedure: blood analysis

INTERVENTIONS:
Procedure: blood analysis — A single venous blood test will be taken - 4 tubes (hematology, clotting, chemistry, sedimentation rate)

SUMMARY:
The investigators hypothesize that low iron storages protects from and down-grades non-alcoholic fatty liver disease.

The aim of the study is to show the association between the severity of Non-alcoholic fatty liver disease to low iron status.

DETAILED DESCRIPTION:
Patients that will pass a CT scan that includes the abdomen will be asked to participate at our study. These patients will be divided into two groups - with and w/o fatty liver. The severity of fatty liver will be determined using the CT scan (as well as other parameters, such as the size of subcutaneous fat layer). Within 72 hours from the scan, a venous blood test will be taken from the enrolled patients (together with a BMI calculation and a blood pressure measurements). In the blood test we will examine liver functions, iron status etc.

This is a preliminary study that will aid in planning future strategies to treat or even prevent fatty liver (one of the epidemics of our century).

ELIGIBILITY:
Inclusion Criteria:

* age>18
* BMI>25

Exclusion Criteria:

* pregnancy
* unable to sign an informed consent (legally)
* known solid/hematological malignancy
* hemoglobinopathy or myelodysplastic disease (not including G6PD deficiency)
* active or carrier of viral hepatitis
* treated a drug the cause fatty liver (eg. amiodarone, tetracyclin, HAART, steroid treatment > 3 months)
* consumption of > 120g ethanol per week
* primary liver disease (eg. glycogen storage disease)
* CRP>20
* acute intoxication
* surgery in previous 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that will pass a CT scan at our institution. The scan must include the abdomen, with or without any contrast material.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
grade of fatty liver disease | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Barzilai medical center, Ashkelon, Israel